CLINICAL TRIAL: NCT05587933
Title: Ejection Fraction of Normal Gall Bladder on Ultrasonography in Patients With Biliary Colic: Is it a Predictor of Cholecystectomy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Yassien Abd-Elkariem, General surgery resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GB EF biliary colic normal US
Record Dates: First submitted 2022-09-24; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Gall Bladder Pain; Hepatobiliary Iminodiacetic Acid; Acalculous Cholecystitis
MeSH Terms: conditions — Acalculous Cholecystitis | interventions — Cholecystectomy; Parasympatholytics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- operative (Experimental)
  Interventions: Procedure: cholecystectomy; Drug: Antispasmodic

INTERVENTIONS:
Procedure: cholecystectomy — cholecystectomy
Drug: Antispasmodic — Antispasmodic

SUMMARY:
In this study investigators aim to evaluate gallbladder ejection fraction as a predictor for cholecystectomy.

DETAILED DESCRIPTION:
The flow of bile through the biliary system is a complex process that depends on the hormonal environment, digestive phase, and functional response of the gallbladder and sphincter of Oddi to all of these factors. Biliary dyskinesia is a disorder of some component of biliary part of the digestive system in which bile cannot physically flow in the proper direction through the tubular biliary tract which causes biliary colic as defined by Rome IV criteria.

Functional causes of biliary pain, also referred to as biliary dyskinesia, are biliary hypokinesia , biliary hyperkinesia and sphincter of Oddi dysfunction (SOD). The exact pathology of functional biliary colic is still unknown. Reviewing Literature status, There is still some debate about the best method to establish the diagnosis gallbladder dyskinesia and hyperkinesia and whether or not ejection fraction is an accurate predictor of outcome. Which led to difficult.

Biliary dyskinesia is identified through gallbladder ejection fraction (GBEF), which is calculated as the flow of radioactive tracer that is ejected from the gallbladder. A GBEF of <35% is considered dyskinesia and a GBEF of <35% is considered hyperkinesia. Patients considered for CCK-HIDA (cholecystokinin hepatobiliary iminodiacetic acid) are those presenting with functional biliary pain based on the Rome IV criteria. Those who present with atypical pain may not need as HIDA (hepatobiliary iminodiacetic acid) as the presentation may be from other pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 14 years of age
* food-related abdominal pain
* normal gallbladder ultrasound (US)
* GB EF 80% and greater or 35% and less on HIDA scan with CCK injection

Exclusion Criteria:

* Patients younger than 14 years old
* Patients with the positive US defined as the presence of gallstones, gallbladder wall thickening (> 4 mm), pericholecystic fluid, sludge, or polyps
* Normal GB EF

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-25 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of quality of life improvment after cholecystectomy according to ROME IV criteria | 6 months
  abdominal pain, nausea and vomiting